CLINICAL TRIAL: NCT04961151
Title: Working Toward the Advancement of Recovery Using Modulated Therapeutic Hyperthermia (WARMTH) in Sepsis - Pilot
Acronym: WARMTH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Nicholas M Mohr (Other)
Collaborators: Hennepin County Medical Center, Minneapolis (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor-Investigator, Nicholas M Mohr, Professor of Emergency Medicine, Anesthesia Critical Care, and Epidemiology, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H202104263
Record Dates: First submitted 2021-06-25; First posted 2021-07-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Sepsis
Keywords: hyperthermia; fever; sepsis
MeSH Terms: conditions — Sepsis; Hyperthermia; Fever

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conductive Wrap Warming (Experimental): Esophageal warming will be discontinued first
  Interventions: Other: Multimodal therapeutic warming w/ esophageal d/c
- Esophageal Warming (Experimental): Conductive wraps will be discontinued first
  Interventions: Other: Multimodal therapeutic warming w/ conductive d/c

INTERVENTIONS:
Other: Multimodal therapeutic warming w/ esophageal d/c — In order to evaluate the ability to reliably raise patient temperature to a target of 39.0°C, patients will be warmed with forced air warming, surface conductive warming, and esophageal core warming. After 4 hours at target temperature, esophageal warming will be discontinued.
  Arms: Conductive Wrap Warming
Other: Multimodal therapeutic warming w/ conductive d/c — In order to evaluate the ability to reliably raise patient temperature to a target of 39.0°C, patients will be warmed with forced air warming, surface conductive warming, and esophageal core warming. After 4 hours at target temperature, conductive warming will be discontinued.
  Arms: Esophageal Warming

SUMMARY:
The purpose of this pilot study is to demonstrate the ability to warm critically ill patients with sepsis to a target temperature of 39°C

DETAILED DESCRIPTION:
Participants with sepsis and without fever will be warmed with surface (forced air and conductive wraps) and core (esophageal) warming, and will have the warming devices placed in the ICU. The warming devices will remain in place until the study is completed (36 hours). The heat exchangers will be set to attain a patient target temperature of 39°C as rapidly as possible, after which the forced-air (non-servo) system will be removed, and the conductive system heat exchanger (powering the water blankets and esophageal device, both of which are servo-controlled) will be set to maintain patient temperature at 39°C for the duration of the study period.

Once goal temperature has been achieved for 2 consecutive hours, the forced air warming device will be discontinued. Patients will be randomized at this point to Group 1, in which esophageal warming will be discontinued first or to Group 2, in which external conductive warming will be discontinued first.

All patients will have usual standard of care labs, vital signs, and imaging for patients undergoing mechanical ventilation in the ICU. For the duration of the 36-hour intervention, patient vital signs, including blood pressure, heart rate, respiratory rate, and vasopressor requirements will be monitored and recorded every 6 hours. Core temperature will be measured and recorded hourly.

Patient's clinical status and outcome will be reviewed in the medical chart 7 days after study completion.

ELIGIBILITY:
Inclusion Criteria:

* Patients above the age of 18 years old.
* Patients with sepsis diagnosed within 48 hours of enrollment. For the purpose of this protocol, sepsis onset is defined as administration of intravenous antibiotics in a patient that the treating critical care physician feels is ill from sepsis.
* All qualifying patients must have a sequential organ failure assessment (SOFA) score of 2 or greater at the time of enrollment.
* Patients requiring mechanical ventilation with an expected duration of mechanical ventilation of >= 2 days.
* Patient maximum baseline documented temperature (within previous 24 hours) < 38.3°C.

Exclusion Criteria:

* Patients without legally authorized representative able to provide informed consent.
* Patients with contraindication to core warming using an esophageal core warming device, surface warming using conductive heat transfer, and forced air warmer.
* Patients known to be pregnant.
* Patients with <40 kg of body mass.
* Patients with comfort care only status.
* Patients with contraindications to hyperthermia treatment (acute stroke, acute traumatic brain injury, acute spinal cord injury, post-cardiac arrest, multiple sclerosis, or sickle cell disease).
* Expected continuous dialysis within 48 hours after enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of warming critically ill patients with sepsis using a multimodal sepsis warming protocol. | 36 hours
  Our primary outcome is the proportion of patients who achieve goal temperature within 6 hours of starting warming. After discontinuing devices, we will monitor the proportion of participants who remain at the goal temperature.
  Warming will be performed using standard technique per instructions for use for the surface warming wraps, esophageal heat transfer device, and forced air warming device. The heat exchanger will be set to a target patient temperature of 39°C, with patient temperature measured via temperature sensing Foley catheter or rectal temperature sensor. Feedback (servo) control is provided by the heat exchanger (Blanketrol III, Gentherm Medical, Cincinnati, OH), such that the water temperature flow through the warming devices is adjusted automatically to enable attainment of the target temperature. Forced air warming will be used until goal temperature is reached for at least 2 hours, then other devices will be used to maintain temperature.

SECONDARY OUTCOMES:
Determine the rate of temperature change of patients undergoing a sepsis warming protocol. | 36 hours
  Participants will be initiated on a warming protocol with forced air warming, surface conductive, and esophageal core warming with the target temperature of 39°C. Patient temperature measurement will be collected hourly during the study period (36 hours).
Determine the ability of conductive heat wraps vs. conductive esophageal device to maintain therapeutic hyperthermia | 36 hours
  Once goal temperature has been achieved for 2 consecutive hours, the forced air warming device will be discontinued. Participants will be randomized at this point to Group 1, in which esophageal warming will be discontinued first or to Group 2, in which external conductive warming will be discontinued first.
  Once goal temperature has been achieved for 4 consecutive hours after discontinuation of the forced air warming device, the second device will be discontinued. If patient body temperature drops below goal temperature, the second warming device will be restarted to maintain temperature.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Mohr, MD, Principal Investigator — University of Iowa
Locations (3):
- United States (3):
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No